CLINICAL TRIAL: NCT03204487
Title: An Open, Non-randomized Study on the Effect of Changing From Preserved Prostaglandin Formulations to Preservative Free Tafluprost (Saflutan® Augentropfen) in Patients With Ocular Hypertension or Primary Open Angle Glaucoma on Tear Film Thickness
Brief Title: A Study on the Effect of Changing From Preserved Prostaglandin Formulations to Preservative Free Tafluprost on Tear Film Thickness
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ordination Dr. Hommer (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HOM1-2015
Record Dates: First submitted 2017-06-23; First posted 2017-07-02 (Actual); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Glaucoma, Open-Angle; Ocular Hypertension
Keywords: tear film thickness; ocular surface disease; OCT
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — tafluprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with glaucoma or ocular hypertension (Experimental)
  Interventions: Drug: Tafluprost 15µg/ml

INTERVENTIONS:
Drug: Tafluprost 15µg/ml — Tafluprost 15µg/ml (Saflutan® 15 microgram/ml Augentropfen im Einzeldosisbehältnis, Merck Sharp & Dohme, Wien)

SUMMARY:
Studies have shown that ocular surface disease (OSD) is common among patients with glaucoma with a prevalence of 50% or more. The percentage of affected patients appears to increase with increasing number of topical anti-glaucoma products instilled. Both pre-clinical and clinical work has indicated that the preservatives used in anti-glaucoma drops, particularly benzalkonium chloride, are mainly responsible for this detrimental effect. As such more and more anti-glaucoma drugs without preservatives entered the market.

To prove that switching from preserved to unpreserved antiglaucoma medication improves the signs and symptom of OSD is, however, not easy. This is on the one hand related to the physiological variability of these parameters over time and on the other hand to the poor association between signs and symptoms. Recently, a new method for measuring tear film thickness (TFT) using ultra-high resolution optical coherence tomography (OCT) has been introduced. Using this method, it has been shown that there is a correlation between reduced TFT and OSD symptoms. In the present study, it is hypothesized that changing patients who are on preserved prostaglandin formulations to preservative free tafluprost may be associated with an increase in TFT.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged over 18 years
* Diagnosed primary open angle glaucoma treated with preserved prostaglandins for at least 6 months OR
* Patients with ocular hypertension treated with preserved prostaglandins for at least 6 months
* IOP ≤ 21 mmHg in the study eye at the screening examination (under treatment)
* Mean TFT at the screening visit ≤ 6µm in the study eye
* At least 2 symptoms of dry eye syndrome in the study eye (itching, stinging, blurred vision, foreign body sensation, debris, conjunctival redness) since at least one month
* Tear break up time ≤ 10sec

Exclusion Criteria:

* Participation in a clinical trial in the 3 weeks before the screening visit
* Severe visual field loss as defined as an MD of -15 or worse in the study eye
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* Presence or history of a severe medical condition that will interfere with the study aim as judged by the clinical investigator
* Sjögren's syndrome
* Stevens-Johnson syndrome
* Presence or history of a severe ocular condition that will interfere with the study aim as judged by the clinical investigator
* Presence or history of allergic conjunctivitis
* Treatment with corticosteroids in the 4 weeks preceding the study
* Wearing of contact lenses
* Topical treatment with any ophthalmic drug in the 4 weeks preceding the study except glaucoma medication or topical lubricants
* Ocular infection
* Ocular surgery in the 6 months preceding the study (except laser trabeculoplasty)
* Pregnancy, planned pregnancy or lactating
* Contraindication against the use of topical prostaglandin therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-05-10 (Actual); Primary Completion 2017-04-25 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Tear film thickness | Change from baseline tear film thickness at 4 and 12 weeks
  Measurement of tear film thickness using OCT

SECONDARY OUTCOMES:
Intraocular pressure (IOP) | Change from baseline IOP at 4 and 12 weeks
  Measurement of IOP using Goldmann applanation tonometry
Ocular Surface Disease Index (OSDI) | Change from baseline OSDI at 4 and 12 weeks
  Subjective symptom questionnaire
Dry-Eye Related Quality of Life Score (DEQS) | Change from baseline DEQS at 4 and 12 weeks
  Subjective symptom questionnaire
Tear Break Up Time (BUT) | Change from baseline BUT at 4 and 12 weeks
  Assessment of BUT in seconds using fluorescein eye drops at the slit lamp.
Schirmer Test 1 | Change from Schirmer Test 1 at 4 and 12 weeks
  Wetting of Schirmer test strips within 5 minutes without topical anaesthesia.
Tear film osmolarity | Change from baseline tear film osmolarity at 4 and 12 weeks
  Tear film osmolarity will be assessed using the TearLab Osmolarity Test.
Corneal fluorescein staining | Change from baseline corneal fluorescein staining at 4 and 12 weeks
  Corneal fluorescein staining will be assessed after instillation of fluorescein eye drops at the slit lamp.

CONTACTS AND LOCATIONS:
Locations (1):
- Ordination Dr. Hommer, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No